CLINICAL TRIAL: NCT02467023
Title: Persistent Inflammation, Immunosuppression and Catabolism Syndrome (PICS): A New Horizon for Surgical Critical Care: Project 4B: Lower Extremity Strength Training in ICU Patients
Brief Title: Project 4B: Lower Extremity Strength Training in ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201500109 -N; P50GM111152-01 (NIH)
Record Dates: First submitted 2015-05-19; First posted 2015-06-09 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Sepsis
Keywords: chronic critical illness; strength training; exercise; sepsis; mechanical ventilation
MeSH Terms: conditions — Sepsis; Motor Activity | interventions — Lidocaine; Biopsy; Midazolam; Fentanyl; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- effective muscle stimulation group (Experimental): Subjects in this arm will be in the study for up to 28 days or until discharge from the ICU. They will receive lower extremity muscle stimulation with Niveus medical stimulator, multiple measurement of maximal isometric twitch strength, muscle biopsy with muscle biopsy medication fentanyl, muscle biopsy medication versed, muscle biopsy medication lidocaine, and blood and urine sampling.
  Interventions: Device: Muscle stimulation with Niveus medical stimulator; Device: measurement of maximal isometric twitch strength; Procedure: Muscle Biopsy; Drug: Muscle Biopsy Medication: Lidocaine; Drug: Muscle Biopsy Medication: Versed; Drug: Muscle Biopsy Medication: Fentanyl; Other: Blood and Urine Sampling
- ineffective muscle stimulation group (Active Comparator): Subjects assigned to this arm will be studied for up to 28 days or until discharge and will receive a sham muscle stimulation with Niveus medical stimulator, multiple measurement of maximal isometric twitch strength blood and urine samples, and a muscle biopsy sample with muscle biopsy medication fentanyl, muscle biopsy medication versed, and muscle biopsy medication lidocaine.
  Interventions: Device: measurement of maximal isometric twitch strength; Procedure: Muscle Biopsy; Drug: Muscle Biopsy Medication: Lidocaine; Drug: Muscle Biopsy Medication: Versed; Drug: Muscle Biopsy Medication: Fentanyl; Other: Blood and Urine Sampling; Device: ineffective muscle stimulation

INTERVENTIONS:
Device: Muscle stimulation with Niveus medical stimulator — Subjects will be treated five days per week, for 30 minutes each session. Muscle stimulation will be conducted for four seconds every 15 seconds, thus the subjects will undergo four stimulations per minute. Muscle stimulation will be adjusted until there is a visible or palpable bilateral quadriceps contraction.
  Arms: effective muscle stimulation group
Device: measurement of maximal isometric twitch strength — Quadriceps strength will be measured on the initial day of study approximately every seven days thereafter and on the final day of study participation. For this measurement, patients will remain supine in their bed and the dominant leg will be placed on a frame that will hold the knee at a 60° angle. A cuff will be placed around the ankle and connected to an electronic dynamometer that will record the force generated during the stimulation. The muscle will be stimulated to contract with magnetic stimulators placed over the body of the quadriceps muscle and stimulated at 100% of power output.
Procedure: Muscle Biopsy — This procedure will be done at the end of participation in the study.The biopsy will be performed with a sterile needle, which will be inserted through the skin. A skin incision (approximately 1/4" long) will be made in order to insert the needle. The biopsy procedure yields two small pieces of muscle tissue (200 mg total), each about half the size of the eraser on a pencil. After the biopsy is taken, the incision will be closed using a steri-strip bandage (no stitches are required), and a sterile dressing will be placed over the site to reduce the risk of bleeding.
Drug: Muscle Biopsy Medication: Lidocaine — Biopsy samples will be obtained under local anesthesia (up to 20 milliliters of 1% Lidocaine administered subcutaneously). Lidocaine, a drug to numb your pain will be injected into the skin and muscle tissue. The injection of the numbing medication will be slightly painful and is similar to receiving a shot into your arm for a vaccination. This medication numbs the skin and muscle so that you do not feel pain when the biopsy is obtained.
  Other Names: Lidocaine for biopsy
Drug: Muscle Biopsy Medication: Versed — Prior to starting the muscle biopsy, you can receive a drug, Versed, to help you relax during the procedure. 1-2 milligrams of Versed will be administered intravenously (in the vein) through an existing peripheral or central intravenous catheter. This procedure drug is given as needed and can be repeated one time as needed.
  Other Names: Versed for biopsy
Drug: Muscle Biopsy Medication: Fentanyl — Prior to starting the muscle biopsy, you can receive a drug, Fentanyl, to make you more comfortable during the procedure. 50-100 micrograms of Fentanyl will be administered intravenously (in the vein) through an existing peripheral or central intravenous catheter. This procedure drug is given as needed and can be repeated one time as needed.
  Other Names: Fentanyl for biopsy
Other: Blood and Urine Sampling — Blood and urine samples will be obtained and examined for markers inflammation and muscle catabolism. Sampling will occur at time of entry into study, and then once every 2-4 days and on the final day of participation or the last day of study (day 28). Peripheral blood will be collected from an existing venous line, or by venipuncture, if required. Urine will be collected from an existing catheter or if the patient is able to void on their own then we will provide a specimen cup. There will be no more than 14 ml of blood drawn at any given time point and a collection of 15 ml of urine at each time point.
Device: ineffective muscle stimulation — An investigator will perform range of motion on both legs, five days per week. The range of motion activity will include the investigator helping you bend and straighten each knee approximately 12 times. Rotation of the leg at the hip will also be performed by bending your knee and gently rotating your upper leg in a clockwise and counterclockwise motion. The range of motion will be performed on each leg and repeated five days per week.
  Arms: ineffective muscle stimulation group

SUMMARY:
The purpose of this research study is to see if electrical stimulation of the leg muscles will improve strength in patients receiving mechanical ventilation in the intensive care unit (ICU). ICU care frequently results in chronically critically ill (CCI) patients. Some CCI patients develop persistent inflammation/immunosuppression and catabolism syndrome (PICS), and they have morbid long-term outcomes. CCI patients with PICS often develop severe limb muscle atrophy, weakness and accelerated protein catabolism. Limb muscle dysfunction in PICS is due to many factors including sepsis/inflammation, proteolysis, apoptosis, and inactivity. Despite the seriousness of limb muscle weakness in CCI patients receiving mechanical ventilation, little is known about exercise strategies to treat this problem. There is limited knowledge about how strength training impacts inflammation and catabolism in CCI patients. In addition, an assessment of the effect of exercise on markers of inflammation and protein catabolism on muscle samples obtained with biopsy techniques and venous blood samples will be performed. This project will further understanding of how treating CCI-related muscle weakness with strength training cannot only improve muscle function, but also potentially blunt the inflammation and catabolism of PICS.

DETAILED DESCRIPTION:
As a participant in the study, the following will take place: Assignment to study groups: a random assignment will be done to one of two groups by a list generated by a computer program, much like flipping a coin. One group of subjects will be assigned to an effective muscle stimulation group and the second group will be assigned to a group that will receive ineffective stimulation (Control or Sham). Muscle stimulation will be performed with a Niveus medical stimulator on both quadriceps muscle groups for 30 minutes, five days per week. The stimulator will be individually adjusted in terms of intensity of stimulation to elicit a visible or palpable quadriceps muscle contraction. Four contractions per minute will be performed for a total of approximately 120 contractions per 30 minute treatment. Isometric Muscle strength testing: All subjects will undergo isometric muscle strength testing. Maximal isometric twitch strength will be measured by placing the subjects' dominant leg in a frame that will hold the knee at 60°. A cuff will be placed around the patient's ankle and will be connected to an electronic dynamometer with the cable. A magnetic nerve stimulator will be used over the body of the quadriceps muscle to stimulate the muscle.

ELIGIBILITY:
Inclusion criteria

1. Presence in the surgery or trauma ICU,
2. age of ≥18 years,
3. received MV for 3 day and expected to survive ICU stay,
4. ability to obtain informed consent from patient or legally authorized representative,
5. approval of an ICU attending for patient to participate.

Exclusion criteria

1. Have an uncontrollable source of sepsis (e.g., irreversible disease state, unresectable dead bowel),
2. are receiving "comfort care" or have advanced care directives limiting resuscitative efforts,
3. have an implanted electronic device (pacemaker/defibrillator/insulin pump, etc.)
4. have known HIV infection with CD4 count < 200 cells/mm3,
5. are organ transplant recipients on immunosuppressive agent(s),
6. have a known pregnancy,
7. history of stroke with weakness,
8. Inability to walk without assistance prior to ICU admission (excluding the use of cane or walker)
9. lower-extremity amputations, rheumatic or severe osteoarthritis of any joint in the lower extremity,
10. Unrepaired hip fracture, unstable cervical spine or other bone diseases
11. arterial or venous insufficiency in the lower extremity,
12. have prior arrangements to be transferred to other facilities before 28 days of treatment,
13. have an unstable or "difficult airway" at 14 days of ICU care, predicted to last for more than 72 hours,
14. are on vasopressor or vasodilatory agents as a continuous infusion at more than a "renal dose,"
15. have severe cardiac dysrhythmias,
16. have acute coronary syndrome,
17. have pulmonary contraindications (pneumo/hemothorax, flail chest),
18. have persistent surgical problems in the post-operative period (serious postoperative bleeding, wound dehiscence, etc.)-when and if these problems resolve and the patient meets other entry criteria, they will be eligible to be recruited for participation,
19. have active neuromuscular diseases that would prevent or interfere with responding to strength training (e.g., amyotrophic lateral sclerosis, multiple sclerosis, myasthenia gravis, polymyositis, muscular dystrophy or other dystrophies and myopathies), and
20. Allergic to lidocaine
21. High risk of bleeding secondary to organic conditions or medication
22. Any anatomical difficulty obtaining biopsy (such a being very overweight)
23. CPR on admission
24. Full dose anticoagulation therapy (ex. Heparin infusion, full anticoagulation dose enoxaparin, Coumadin/Warfarin/Jantoven/Marevan/Waran, and Argatroban).
25. Patient on antiplatelet therapy and medicine such as Plavix (also known as Clopidogrel, Clopilet, and Ceruvin), Aggrenox (also known as aspirin with Dipyridamol), Ticlid (also known as ticlopidine), Agrylin or Xagrid (also known as Anagrelide). Of note, aspirin is not an exclusion criteria, as long as that is the only anti-platelet medication the patient is receiving. In addition, other non steroidal anti-inflammatory agents-NSAIDS (Ibuprofen, Naproxen, Indomethicin or other anti-inflammatories) are not a contraindication to the muscle biopsy procedure and
26. any other factor in the investigators' judgment that would unnecessarily increase the risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07-07 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Isometric muscle twitch force measured at the start of the study, approximately every seven days thereafter and final day of study. | Change from days 1, 7, 14, 21, and 28
  Measurement of maximal isometric strength will be done by using a dynamometer.
Change in inflammatory markers on days 1, 7, 14, 21, and 28. | Change from days 1, 7, 14, 21, and 28
  blood and urine will be tested for the markers of inflammation. The following will be tested: (IL)-1β, IL-6, IL-8, IL-10, IL-12, (TNF)α, (IFN)γ, (MCP)-1, (IP)10, (SDF)-1, (MIP)1α, (HMG)B1, procalcitonin, and (CRP).
Change in immunosuppressive markers on days 1, 7, 14, 21, and 28. | Change from days 1, 7, 14, 21, and 28
  blood and urine will be tested for the markers of immunosuppression. The following will be tested: MDSC phenotype (HLA-DRlow)

SECONDARY OUTCOMES:
Measurement of key proteins of mitochondrial function using immunohistochemistry and Western blotting | Measurement on day 28
  Quadriceps muscle samples will be obtained with percutaneous biopsies following training. Muscle fiber cross-sectional area, myosin heavy chain composition, and changes in atrophy-specific proteins will be assessed using immunohistochemistry and Western blotting, respectively. High-resolution respirometry on permeabilized muscle fibers will be used to measure changes in mitochondrial O2 consumption and muscle bioenergetics. In addition, we will measure key proteins of mitochondrial function and biogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Martin, PhD, PT, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Hospital at the University of Florida, Gainesville, Florida, United States